CLINICAL TRIAL: NCT01930149
Title: Reducing Disparities in Primary Prevention of Cardiovascular Disease: Promoting Cholesterol Screening
Brief Title: Promoting Cholesterol Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stephen Persell, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1PO1HS021141-01-Project 2B; 1P01HS021141-01 (NIH)
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Cardiovascular Diseases; Lipid Testing; Primary Prevention of Cardiovascular Disease
Keywords: Cholesterol screening; High cholesterol; Cardiovascular disease; Statin treatment
MeSH Terms: conditions — Cardiovascular Diseases; Hypercholesterolemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mailed patient outreach intervention (Experimental): Participants randomized to this arm will receive mailed letter from health center that encourages cholesterol testing and describes the steps necessary to obtain the test at the patient's care site. Clinic staff will facilitate the ordering of tests for patients who may not have an office visit.
  Interventions: Behavioral: Mailed patient outreach intervention
- Usual Care Control Group (No Intervention): Participants randomized to this arm will receive usual care.

INTERVENTIONS:
Behavioral: Mailed patient outreach intervention — This study's intervention is a mailed outreach letter from the health center that encourages cholesterol testing and describes the steps necessary to obtain the test at the patient's care site. Clinic staff will facilitate the ordering of tests for patients who may not have an office visit.
  Arms: Mailed patient outreach intervention

SUMMARY:
Cholesterol screening is an important prerequisite for cardiovascular disease (CVD) risk assessment. Cholesterol screening is recommended by the United States Preventive Services Task Force (USPSTF). Since reminder systems have been shown to modestly improve the rates of preventive services, including in safety net settings, we will implement patient-directed reminders to health center patients who meet our eligibility criteria.

The aim of this study is to determine if a mailed outreach message and facilitated ordering of screening lipid tests increases cholesterol screening test completion within 3 months among federally qualified community health center patients who are eligible for screening compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patient at participating health center
* At least 1 visit to clinic in the prior 12 months
* No total cholesterol and high-density lipoprotein cholesterol result recorded in the electronic health record in the past 5 years
* No cholesterol screening order placed within the previous 3 months
* Men 35-75 years old, or women 45-75 years old who also have one of the following: hypertension, obesity, or current smoking

Exclusion Criteria:

* Previously diagnosed cardiovascular disease, peripheral arterial disease or diabetes mellitus
* Statin on active medication list
* Preferred language other than English or Spanish

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Completion of total cholesterol and HDL cholesterol test or full lipid panel | within 3 months of outreach
  Primary outcome will be completion of total cholesterol and HDL cholesterol test or a full lipid panel recorded within GE Centricity electronic health record at the patient's clinical site.

SECONDARY OUTCOMES:
Statin prescription | within 3 months of outreach
  Secondary outcome is prescription of a statin as assessed by automated electronic queries of electronic health record.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Persell, MD, MPH, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - North Country Health Care, Flagstaff, Arizona
  - Near North Health Service Corporation, Chicago, Illinois
  - Heartland Health Outreach, Chicago, Illinois